CLINICAL TRIAL: NCT06099457
Title: SIBTime: Media-enhanced Technology for Promoting the Behavioral Health and Family Relationships of Typically Developing Young Siblings
Brief Title: SIBTime Phase II: Web Application for Typically Developing Siblings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD015947-02; 2R44MD015947-02 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Early Life Stress
Keywords: Siblings; Disability; Health concern
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: One intervention and two arms (intervention and waitlist control group, treatment-as-usual).
  Randomly assign 80 parent participants to a treatment condition and 80 to waitlist control group, treatment-as-usual. Conduct an 8-week intervention among the treatment condition participants. At the conclusion of post-intervention testing, deliver the SIBTime intervention to the treatment-as-usual condition participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Sibtime web-based intervention.
  Interventions: Behavioral: SIB-Time web-application tool
- Control (No Intervention): Business as usual.

INTERVENTIONS:
Behavioral: SIB-Time web-application tool — Parent-child dyads will use the SIBTime app in an 8-week intervention to test its relevance, acceptability, cultural appropriateness, and potential for efficacy.
  Arms: Treatment

SUMMARY:
Most of the over 32.7 million people in the U.S. who have special health, developmental, and mental health concerns have typically developing (TD) brothers and sisters who share high levels of involvement in their sibling's lives. Disability and health agencies lack effective tools to support the information and support needs of TD siblings and their families, in particular for ethnic minority and rural families. The aims of this proposal are to complete development and evaluation of the dual language SIBTime app, designed to build parents' and children's knowledge, skills, and engaging family routines to nurture TD siblings' (ages 3-6) social-emotional health and well-being.

DETAILED DESCRIPTION:
An 8-week RCT will be conducted to evaluate the full-scale SIBTime program in a sufficiently powered randomized controlled trial evaluation (sample size = 160 parent/child dyads). SIBTime will be assessed in terms of its relevance, acceptability, cultural appropriateness, and efficacy. Participants will complete measures pre- and post- intervention selected to detect changes in parenting stress and adjustment, parent-child relationship, parents' self-efficacy and frequency of engagement in the targeted parenting strategies, and TD sibling behavior and adjustment. Information will also be collected on family demographics, consumer satisfaction, usability ratings, usage metrics, and recommendations for modifications to the program.

ELIGIBILITY:
Criteria:

Inclusion criteria:

1. Parent of a child with a disability and a typically developing child aged 3-6
2. Has a smartphone or tablet
3. Speaks English or Spanish

Exclusion criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Child-Parent Relationship Scale - Short Form | Baseline and Week 9
  The Child-Parent Relationship Scale - Short Form (CPRS-SF; Driscoll & Pianta, 2011) is used to measure the degree of closeness and conflict in the parent-child relationship. The CPRS-SF is comprised of 15 parent-report items that ask the parent for their assessment of the child-parent relationship, the child's emotional stance toward the parent, and the parent's feelings toward the child. Items are answered on a 5-point "Definitely does not apply" to "Definitely applies" scale. Two subscales are derived: Conflicts and Positive Aspects/Closeness. Both subscales are measured by 7 items, which are averaged together; average scores range from 1 to 5. For the Conflicts subscale, higher scores indicate worse outcomes; for the Closeness subscale, higher scores indicate better outcomes. The CPRS-SF has been validated with parents of preschoolers and first graders, and shows good internal consistency with acceptable Cronbach alphas (.64-.84).
Parental Stress Scale | Baseline and Week 9
  The Parental Stress Scale (PSS; Berry and Jones, 1995) is used to measure parents' stress level. The PSS is comprised of 18 items that ask about positive (emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. Respondents answer on a 5-point Likert "Strongly agree" to "Strongly disagree" scale in terms of their typical relationship with their child(ren). Summed scores range from 18 to 90, with higher scores indicating worse outcomes. The PSS shows good internal consistency, test-retest reliability, discriminant validity, and construct validity (Berry & Jones, 1995). It has been validated across cultures and languages (Louie, Cromer, & Berry, 2017), with families of TD children, and with families of children with emotional/ behavioral problems, developmental disabilities (Berry & Jones, 1995), and chronic health conditions (Zelman & Ferro, 2018).
Self-Efficacy for Parenting Tasks Index - Toddler Scale | Baseline and Week 9
  The Self-Efficacy for Parenting Tasks Index - Toddler Scale (SEPTI-TS; Coleman & Karraker, 2003) is used to measure parents' self-efficacy for a broad range of parenting tasks involved in ensuring the wellbeing of the target TD child. Four subscales of the SEPTI will be used: Emotional Availability (7 items), Nurturance/Valuing/ Empathetic Responsiveness (8 items), Play (7 items), and Teaching (9 items). Items are answered on a 6-point Likert response scale (1= Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating lower self-efficacy (worse outcome). The SEPTI-TS shows good internal consistency, construct validity, discriminant validity, and sensitivity to change.
Engagement in Target Activities with Child - Frequency Subscale | Baseline and Week 9
  The frequency of parents' engagement in the parenting practices targeted by the intervention is measured via the Engagement in Target Activities with Child measure, Frequency subscale. Created for this study, these 22 items ask parents to report the frequency with which they have engaged in target parenting practices in the past month; parents report their frequency on a 7-point scale ("Never in the past month" to "6 or more times per day"). Averaged scores range from 0 to 6, with higher scores indicating more frequent parental engagement in the target activities (better outcome).
Engagement in Program-Targeted Activities with Child - Parents' Self-Efficacy Subscale | Baseline and Week 9
  Parents' self-efficacy for engaging in the parenting practices targeted by the intervention is measured via the Engagement in Target Activities with Child measure, Parents' Self-Efficacy subscale. Created for this study, these 22 items ask parents to rate how confident they are that they know how to do a series of parenting practices targeted by the program, on a scale of 0 to 4 (0 = I don't know how to do this at all, 4 = I know how to do this very well). Averaged scores range from 0 to 4, with higher scores indicating greater parental self-efficacy that they know how to do the target activities (better outcome).
Parents' Rating of their Own Program-Targeted Behaviors | Baseline and Week 9
  Parents' perception of their TD child's engagement in program-targeted behaviors is measured with parents' rating on 4 child behaviors targeted by the program, and one item asking about the child's general adjustment to their sibling's disability/illness. Created for this study, 4 of the items ask parents to report the frequency with which their TD child has engaged in target behaviors in the past month; parents report their frequency on a 7-point scale ("Never in the past month" to "6 or more times per day"). Averaged scores range from 0 to 6, with higher scores indicating more frequent child engagement in the target activities (better outcome). The 5th item asks parents how satisfied they are with how well their TD child is doing, as a sibling of a child with a disability or health concern. Parents respond on a scale of 1 to 10, with 1 = Not at all satisfied and 10 = Very satisfied.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) -- Ages 3 to 4 | Baseline and Week 9
  Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) is used to measure the TD child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior that can be completed in about 5 minutes. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior. Respondents answer on a 3-point (from 0 to 2) "Not true" to "Certainly true" scale. For problem behavior subscales, higher scores indicate worse adjustment; for the prosocial behavior scale, higher scores indicate better adjustment. The SDQ shows good construct and discriminant validity and is sensitive to both child internalizing and externalizing behavior.
System Usability Scale (SUS) | Week 9 only
  Skill usability is measured with the System Usability Scale (SUS), a commonly used 10-item scale that measures subjective perceptions of usability. Items are answered on a 5-point scale (0=Strongly disagree; 4=Strongly agree); scores on the scale are summed and multiplied by 2.5, such that they range from 0 to 100, with higher scores indicating better usability. The SUS has been normed, and scoring produces an overall usability "grade" (Brooke, 1996; Sauro, 2011). This measure is obtained from only from treatment participants only at post-test.
Parent Satisfaction | Week 9 only
  Parents' satisfaction with the SibTime app will be measured with 9 items that ask parents to rate, on a 5-point response scale (e.g. 1=Not at all; 5=Very much), the degree to which the SibTime app was helpful to them and to their child, addressed topics important to their family, enjoyable, and their overall satisfaction with the SibTime app. Scores are averaged across items, with higher scores indicating greater satisfaction (better outcomes). This measure will be obtained only from treatment participants only at posttest.
Family usage of the SIBTime program | Week 9 only
  Families' usage of the SIBTime app is measured through usage metrics collected on the back-end database, including whether or not the app is activated, which elements are accessed; frequency and duration of engagements; and points of difficulty or failure. These metrics are collected from users in the treatment condition only.
Commercial Feasibility | Month 21
  Commercial feasibility will be measured with the Practitioner Satisfaction & Program Acceptability measure, 20 items that Advisory Board members and recruitment partners will complete. These items measure SIBTime's acceptability for the target families these practitioners serve, feasibility for use among agencies, and interest in purchasing and adopting SIBTime.
Sibling Inventory of Behavior | Baseline and Week 9
  The parent's perceptions of their children's sibling relationship is measured with the Sibling Inventory of Behavior. The instrument (SIB; Schaeffer & Edgerton, 1981; Volling & Blandon, 2003) has 6 subscales: Companionship/Involvement, Empathy/Concern, Teach/Manage/Directiveness, Rivalry, Aggression/Conflict, and Avoidance. The Teach/Mange/Directiveness subscale was not used, and the number of items in the Rivalry scale was reduced from 7 to 5 to reduce length and participant burden. Parents answer on a 5-point Never to Always scale. Average scores range from 1 to 5. For Positive subscales (Companionship/Involvement and Empathy/Concern), higher scores indicate a better relationship; for Negative subscales (Rivalry, Aggression/Conflict, and Avoidance), higher score indicate a worse relationship. Scores can be analyzed at the subscale level, as well as at the composite "Positive" and "Negative" levels.
Parent's Rating of Their Child's Program-Targeted Behaviors | Baseline and Week 9
  Parents' perception of their TD child's engagement in program-targeted behaviors is measured with parents' rating on 4 child behaviors targeted by the program, and one item asking about the child's general adjustment to their sibling's disability/illness. Created for this study, 4 of the items ask parents to report the frequency with which their TD child has engaged in target behaviors in the past month; parents report their frequency on a 7-point scale ("Never in the past month" to "6 or more times per day"). Averaged scores range from 0 to 6, with higher scores indicating more frequent child engagement in the target activities (better outcome). The 5th item asks parents how satisfied they are with how well their TD child is doing, as a sibling of a child with a disability or health concern. Parents respond on a scale of 1 to 10, with 1 = Not at all satisfied and 10 = Very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Marquez, BA, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- David R Smith, Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Driscoll, K., & Pianta, R. C. (2011). Mothers' and fathers' perceptions of conflict and closeness in parent-child relationships during early childhood. Journal of Early Childhood and Infant Psychology, 7, 1-24.
- [Background] Berry, J. O., & Jones, W. H. (1995). The Parental Stress Scale: Initial psychometric evidence. Journal of Social and Personal Relationship, 12(3), 463-472.
- [Background] Louie, A. D., Cromer, L. D., & Berry, J. O. (2017). Assessing parenting stress: Review of the use and interpretation of the Parental Stress Scale. The Family Journal, 25(4), 359-367.
- [Background] Zelman, J. J. & Ferro, M. A. (2018). The Parental Stress Scale: Psychometric properties in families of children with chronic health conditions. Family Relations, 67(2), 240-252.
- [Background] Coleman, P. K. & Karraker, K. H. (2003). Maternal self-efficacy beliefs, competence in parenting, and toddlers' behavior and developmental status. Infant Mental Health Journal, 24(2), 126-148.
- [Background] Lobato DJ, Kao BT. Integrated sibling-parent group intervention to improve sibling knowledge and adjustment to chronic illness and disability. J Pediatr Psychol. 2002 Dec;27(8):711-6. doi: 10.1093/jpepsy/27.8.711. PMID 12403861
- [Background] Sahler OJ, Carpenter PJ. Evaluation of a camp program for siblings of children with cancer. Am J Dis Child. 1989 Jun;143(6):690-6. doi: 10.1001/archpedi.1989.02150180068023. PMID 2729214
- [Background] Guite, J., Lobato, D., Kao, B, & Plante, W. (2010). Discordance between sibling and parent reports of the impact of chronic illness and disability on siblings. Children's Health Care, 33(1), 77-92.
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Brooke, J. (1996). SUS: A "quick and dirty" usability scale. In P. W. Jordan, B. Thomas, B. A. Weerdmeester, & A. L. McClelland (Eds.), Usability evaluation in industry. Taylor and Francis.
- [Background] Sauro J. (2011). A practical guide to the System Usability Scale: Background, benchmarks & best practices. Measuring Usability LLC.